CLINICAL TRIAL: NCT01617200
Title: A Multicenter, Double-Blind, Fixed-Dose, Long-Term Extension Trial of the Safety of Asenapine Using Olanzapine as an Active Control in Subjects Diagnosed With Schizophrenia Who Completed Protocol P05688
Brief Title: Long-Term Safety Extension Trial of Asenapine in Schizophrenia Participants Who Completed Protocol P05688 (P05689)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05689; 2010-018408-96 (EudraCT Number)
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — asenapine; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Asenapine 2.5 mg BID (Experimental)
  Interventions: Drug: Asenapine; Drug: Placebo Olanzapine
- Asenapine 5 mg BID (Experimental)
  Interventions: Drug: Asenapine; Drug: Placebo Olanzapine
- Olanzapine 15 mg QD (Active Comparator)
  Interventions: Drug: Placebo Asenapine; Drug: Olanzapine; Drug: Placebo Olanzapine
- Placebo switched to Asenapine 2.5 mg BID (Experimental)
  Interventions: Drug: Asenapine; Drug: Placebo Olanzapine

INTERVENTIONS:
Drug: Asenapine — 2.5 mg or 5 mg fast dissolving active asenapine tablets administered sublingually, same number of tablets are taken in the morning and the evening
  Other Names: Saphris®; SCH 900274; Org 5222; Sycrest®
  Arms: Asenapine 2.5 mg BID; Asenapine 5 mg BID; Placebo switched to Asenapine 2.5 mg BID
Drug: Placebo Asenapine — 2.5 mg or 5 mg fast dissolving placebo asenapine tablets administered sublingually, same number of tablets are taken in the morning and the evening
  Arms: Olanzapine 15 mg QD
Drug: Olanzapine — 15 mg film-coated active olanzapine tablets administered orally QD. The time of the active olanzapine dose (either morning or evening) is not disclosed in order to preserve blinding.
  Other Names: Zyprexa
  Arms: Olanzapine 15 mg QD
Drug: Placebo Olanzapine — 15 mg film-coated placebo olanzapine tablets administered orally QD. The time of the active olanzapine dose (either morning or evening) is not disclosed in order to preserve blinding.

SUMMARY:
Participants who have completed the 6-week trial P05688 can be screened for eligibility for this 26-week extension study in which they will continue treatment. The purpose of this trial is to evaluate the long-term safety of 2.5 and 5 mg asenapine administered sublingually twice daily (BID) in schizophrenia participants. Olanzapine administered 15 mg orally once daily (QD) is used as an active control.

ELIGIBILITY:
Inclusion Criteria:

* Completed the short-term trial P05688, and judged by the investigator likely to benefit from continued treatment

Exclusion Criteria:

* Occurrence(s) of an adverse event or other clinically significant finding(s) in the short-term trial P05688 that would prohibit the participant's continuation into the long-term extension
* Clinical Global Impression-Severity of Illness (CGI-S) score of ≥6 (severely psychotic) at Baseline
* Newly diagnosed or discovered psychiatric condition that would have excluded the participant from participation in the short-term trial P05688

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in Weight From Baseline to Day 182 | Baseline (Day -1 of Short Term Trial) to Day 182 (Long-Term Extension)

CONTACTS AND LOCATIONS:
Locations (1):
- Forest Investigative Site 2001, Austin, Texas, United States